CLINICAL TRIAL: NCT07308041
Title: An Open, Single Arm, Single-center, Phase 1 Trial Investigating the Effect of 7-days-repeated Administration of Linaprazan Glurate on the Pharmacokinetics of Repeated Doses of Amoxicillin in Healthy Participants
Brief Title: A Study to Investigate the Effect of Linaprazan Glurate on the Pharmacokinetics of Amoxicillin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cinclus Pharma Holding AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CX842B2111
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Drug Interaction; GERD (Gastroesophageal Reflux Disease); Safety, and Tolerability
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Drug Interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Linaprazan glurate (Experimental): Oral administration for seven (7) days.
  Interventions: Drug: Drug Drug Interaction

INTERVENTIONS:
Drug: Drug Drug Interaction — The intervention phase consists of 2 periods: in period 1, the pharmacokinetics (PK) of amoxicillin will be evaluated in the absence of linaprazan glurate, in period 2, a potential effect of linaprazan glurate on the PK of amoxicillin will be evaluated as well as the PK of linaprazan glurate following co-administration of amoxicillin.

SUMMARY:
This is an open, single arm, single-center Phase I trial designed to evaluate the effect of seven days repeated oral doses of linaprazan glurate on the pharmacokinetics (PK) of repeated doses of amoxicillin in healthy male and female participants

DETAILED DESCRIPTION:
Participants in the trial will attend three visits to the clinical research unit (CRU) and a telephone follow-up visit.

Eligible participants will be admitted to the CRU in the evening of Day -1 and will remain at the CRU until the morning of Day 2 In the morning of Day 1, after pre-dose assessments, a dose of amoxicillin will be administered followed by 24 hours PK blood sampling for determination of amoxicillin plasma concentrations. Safety will be followed up throughout the 24 hours. In the morning of Day 2, after the 24-hour amoxicillin PK sample and safety assessments, the first linaprazan glurate will be administered to the participants. The participants will then continue to take linaprazan glurate (Day 2 to Day 8).

The participants will be admitted to the CRU in the afternoon of Day 6 and will remain at the CRU until the morning of Day 9. PK samples for determination of linaprazan glurate and linaprazan in plasma will be collected for 24 hours at Day 7. In the morning of Day 8, the participants will be administered a new dose of amoxicillin together with the dose of linaprazan glurate, which will be followed by 24 hours PK sampling for determination of amoxicillin, linaprazan glurate and linaprazan plasma concentrations. The participants will leave the CRU after the 24-hour PK sample and safety assessments.

A final end-of-trial telephone call will take place seven days (±two days) after the final dosing on Day 8.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the trial.
* Healthy male or female participant aged 18 to 64 years, inclusive.
* Body mass index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2 at the time of the screening visit.
* Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values at the time of the screening visit, as judged by the Investigator.
* Prospective participants, as well as their partners, must agree to the contraception requirements described in exclusion criteria 1 and 2.

Exclusion Criteria:

* Female participants of childbearing potential (defined as all participants physiologically capable of becoming pregnant) unless they agree to use one of the following highly effective methods of contraception (failure rate of <1%) from 2 weeks prior to the first dose until the end-of-trial visit:

  * Sterilization of a male partner, defined as vasectomy, at least six months prior to screening.
  * Intra-uterine device (non-hormonal or copper IUD).
  * Double-barrier methods of contraception, i.e., condoms in combination with occlusive cap with contraceptive gel.
* Male participants with a partner of childbearing potential, unless they agree to use one of the following methods of contraception from two weeks prior to the first dose until the end-of-trial visit:

  * Vasectomy at least six months prior to screening.
  * Condoms. Female partners of childbearing potential must then agree to concurrently use a highly effective method of contraception.
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results or the participant's ability to participate in the trial.
* Any clinically significant illness, medical/surgical procedure or trauma within four weeks of the first administration of IMP.
* Positive result for H.pylori antibodies at the time of the screening visit.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Characterization of the PK of amoxicillin following a repeated dose before and after repeated administration of linaprazan glurate (AUC) | Day 1 and Day 8
  Geometric mean ratio Day 8/Day 1 for amoxicillin Area Under the Plasma Concentration vs. Time Curve (AUC)
Characterization of the PK of amoxicillin following a repeated dose before and after repeated administration of linaprazan glurate (Cmax) | Day 1 and Day 8
  Geometric mean ratio Day 8/Day 1 for amoxicillin Cmax
Characterization of the PK of amoxicillin following a repeated dose before and after repeated administration of linaprazan glurate (Tmax) | Day 1 and Day 8
  Amoxicillin Tmax
Characterization of the PK of amoxicillin following a repeated dose before and after repeated administration of linaprazan glurate (CL/F) | Day 1 and Day 8
  Amoxicillin apparent oral clearance (CL/F)

CONTACTS AND LOCATIONS:
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No